CLINICAL TRIAL: NCT00174759
Title: A Double-blind, Randomized Study of Clopidogrel 75 mg/d vs Placebo, on a Background of ASA 75-100 mg/d,in Peripheral Arterial Disease (PAD) Patients Receiving a Unilateral Below Knee Bypass Graft.
Brief Title: CASPAR : Clopidogrel and Acetyl Salicylic Acid in Bypass Surgery for Peripheral ARterial Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C_9253; EudraCT #: 2004-000822-58
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Arterial Occlusive Diseases
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel

SUMMARY:
Primary objective:

To evaluate whether clopidogrel 75 mg o.d. versus placebo (on a background of ASA 75-100 mg/d) will lead to an increased rate of primary patency, limb salvage and survival, in patients receiving a below knee bypass graft for the treatment of PAD.

Secondary objectives:

Comparison, between the two treatment groups, of :

* Primary patency,
* Assisted primary patency,
* Cardiovascular death / myocardial infarction / stroke / any amputation above the ankle.
* Ankle Brachial Pressure Index (ABPI) changes from baseline

ELIGIBILITY:
Inclusion Criteria: A patient is eligible for inclusion in the study 2-4 days after surgery if all the following criteria are fulfilled:

* Informed consent obtained;
* Chronic background treatment with daily ASA, whatever the dose, started at least 4 weeks before surgery. A window of a few days without ASA before surgery is acceptable, according to local practice. Post-randomization use of ASA must be between 75 and 100 mg/day.
* Unilateral below knee bypass graft (i.e. the distal anastomosis is below the level of the knee joint) for atherosclerotic PAD within the previous 4 days;
* Demonstration of initial patency of the index graft by an objective measurement (e.g. intra-operative Doppler scanning, flow measurement, angiography, Duplex scanning) during bypass surgery, or between surgery and the time of randomization;
* No clinical evidence of graft occlusion at time of randomization.

Exclusion criteria :

PAD medical/surgical history

* Onset of PAD symptoms before the age of 40 years
* Non-atherosclerotic vascular disease (e.g. Buerger's disease, popliteal entrapment syndrome)
* Patient receiving aorto-bifemoral, iliac-femoral or crossover (femoral-femoral) grafts, or undergoing peripheral transcutaneous angioplasty (PTA), with or without stenting, during the same surgery.

Medical history related to bleeding risk

* Current active bleeding at surgical site
* Withdrawal of an epidural catheter less than 12 hours before randomization
* Current active bleeding or increased risk of bleeding, such as severe hepatic insufficiency, proliferative diabetic retinopathy, peptic ulceration, bleeding diathesis or coagulopathy
* Peptic ulceration within 12 months of randomization
* Previous or current intracranial hemorrhage or hemorrhagic stroke, or any previous stroke for which the diagnosis of hemorrhagic stroke cannot be excluded
* Any history of severe spontaneous bleeding such as gastrointestinal bleeding, gross hematuria, intraocular bleeding

Other medical conditions

* Previous disabling stroke (severe cerebral deficit such that the patient is bedridden or demented)
* NYHA Class IV heart failure
* Uncontrolled hypertension: Systolic Blood Pressure (SBP) > 180 mm Hg, or Diastolic Blood Pressure (DBP) > 100 mm Hg

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1460 (Estimated)
Dates: Start 2004-09

PRIMARY OUTCOMES:
1st occurrence over the duration of follow-up of : index bypass graft occlusion based on imaging procedure, or graft replacement or endovascular intervention, or amputation above the ankle of the affected limb or death

SECONDARY OUTCOMES:
1st occurrence of any component of following cluster of events : index bypass graft occlusion,any revascularization procedure or amputation. Change in ABPI.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Sagnard, Study Director — Sanofi
Locations (14):
- Sanofi-Aventis, North Ryde, Australia
- Sanofi-Aventis, Vienna, Austria
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Helsinki, Finland
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Budapest, Hungary
- Sanofi-Aventis, Milan, Italy
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Stockholm, Sweden
- Sanofi-Aventis, Meyrin, Switzerland
- Sanofi-Aventis, Guildford, United Kingdom

REFERENCES:
- [Derived] Belch JJ, Dormandy J; CASPAR Writing Committee; Biasi GM, Cairols M, Diehm C, Eikelboom B, Golledge J, Jawien A, Lepantalo M, Norgren L, Hiatt WR, Becquemin JP, Bergqvist D, Clement D, Baumgartner I, Minar E, Stonebridge P, Vermassen F, Matyas L, Leizorovicz A. Results of the randomized, placebo-controlled clopidogrel and acetylsalicylic acid in bypass surgery for peripheral arterial disease (CASPAR) trial. J Vasc Surg. 2010 Oct;52(4):825-33, 833.e1-2. doi: 10.1016/j.jvs.2010.04.027. Epub 2010 Aug 1. PMID 20678878